CLINICAL TRIAL: NCT02310854
Title: Acute Anterior Cruciate Ligament Rupture; RecOnsTruction Or Repair?
Acronym: ROTOR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedisch Centrum Oost Nederland (Other)
Responsible Party: Principal Investigator, Judith olde Heuvel, PhD, Orthopedisch Centrum Oost Nederland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL5011604414
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: anterior cruciate ligament rupture; autograft; reconstruction; orthopedic surgery; dynamic intraligament stabilization
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACL Reconstruction (Active Comparator): Primary reconstructive surgery of ACL with hamstring autograft (All-inside, Arthrex, Napels, Florida, USA)
  Interventions: Procedure: ACL reconstruction
- ACL Repair (Experimental): Primary augmented suture of ACL using Dynamic Intraligament Stabilization (DIS; Mathys Medical Bettlach, Switzerland)
  Interventions: Procedure: ACL Repair

INTERVENTIONS:
Procedure: ACL Repair — augmented suture of acute ACL rupture (<3 weeks after injury)
  Other Names: Dynamic Intraligament Stabilization (DIS); Augmented suture
  Arms: ACL Repair
Procedure: ACL reconstruction — reconstruction hamstring autograft
  Other Names: Primary ACL reconstruction; Autograft hamstring; All-inside
  Arms: ACL Reconstruction

SUMMARY:
To investigate the hypothesis that suture repair of a ruptured vkb, combined with a dynamic intraligamentary stabilization and microfracture of the femoral notch, results in at least equal effectiveness compared with an ACL reconstruction using autologous hamstring in terms of functional recovery one year postoperatively in terms of a patient self-reported outcome related to be able to conduct daily and sporting activities. Secondary, the evaluation of clinical outcomes, self-reported by the patient outcomes, osteoarthritis, rehabilitation time required for return to daily and sporting activities and levels of sporting activity which has returned in patients with status after an ACL rupture and suture repair augmented with a dynamic intraligamentary microfracture and stabilization of the femoral notch in comparison with an anterior cruciate ligament reconstruction with the ipsilateral hamstring graft.

DETAILED DESCRIPTION:
Background of the study:

An anterior cruciate ligament rupture is a serious injury to the knee with high probability of the occurrence of dynamic instability, accompanying lesions and early post-traumatic arthrosis. Despite conservative treatment through rehabilitation or ACL reconstruction surgery not all patients do return to their previous activity levels. Moreover degenerative changes, especially early posttraumatic arthrosis, are not counteracted.

In order to optimize the clinical results after ACL surgery, a renewed interest has emerged in healing the patient's own ruptured ACL after attaching. Literature suggests that with the current innovations in surgical repair techniques of (natural) healing of a ruptured ACL may result in similar clinical outcomes in comparison to the gold standard, the ACL reconstruction. In addition, it may even reduce degenerative changes occur in relation to the gold standard. Moreover, the return to daily activities and sports level seems significantly faster than after ACL reconstruction.

The hypothesis is that a suture (suture repair) of a ruptured ACL, combined with a dynamic intraligamentary stabilization, as well as microfracture of the femoral notch, passes, at least equal efficacy in comparison with an anterior cruciate ligament reconstruction using autologous hamstrings in terms of functional recovery 1 years postoperatively.

The DIS bonding technique will be applied in the current study to surgically repair (suture) the ruptured ACL. DIS is an abbreviation and stands for intraligamentary dynamic stabilization (DIS). DIS has been used in humans and seems to provide a high patient satisfaction, favorable clinical and radiological results. However, to our knowledge, to date, no randomized comparative study has been conducted yet in which the DIS technique is compared with the gold standard, the ACL reconstruction.

Objective of the study:

Primary goal:

Investigate the hypothesis that suture repair of a ruptured vkb, combined with a dynamic intraligamentary stabilization and microfracture of the femoral notch, results in at least equal effectiveness compared with an ACL reconstruction using autologous hamstring in terms of functional recovery one year postoperatively in terms of a patient self-reported outcome related to be able to conduct daily and sporting activities.

Secondary objective:

Evaluation of clinical outcomes, self-reported by the patient outcomes, osteoarthritis, rehabilitation time required for return to daily and sporting activities and levels of sporting activity which has returned in patients with status after an ACL rupture and suture repair augmented with a dynamic intraligamentary microfracture and stabilization of the femoral notch in comparison with an anterior cruciate ligament reconstruction with the ipsilateral hamstring graft.

Study design:

This study is a single center stratified block randomized controlled trial. Patients with ACL rupture, confirmed by an orthopedic surgeon based on the outpatient history and radiographic images, will be randomized into an experimental ('repair' / DIS) group after inclusion and a control (reconstruction, regular care) group. Patients will be stratified on the level of sport/physical active practice, on the basis of the Tegner score. The Tegner score is an evaluative and inventory questionnaire on which the patient indicates the gravity of his work and/or sports activities. A higher score is associated with a higher level of physical strain/activity . On the basis of the Tegner score patients will be stratified into a 'moderate' physically active stratum (group Tegner score 5-6-7) and 'highly' physically active stratum (group Tegner score 8 -9-10). Stratification based on the degree of physical activity is considered to be important because the extent and severity of physical activity/strain in daily life poses a potential (difference) in risk of re-rupture between the two study arms. In order to minimize potential differences in 'exposure' or 'risk of re-rupture' between the two study groups stratification is relevant.Measurements take place at baseline, peri-operative / immediately after surgery, 6 weeks, 3,6,9 months and 1, 2, 5 and 10 years postoperatively.

Study population: (Physically) active patients from 18 untill 30 years, who has visited the outpatient clinic of the orthopedic surgeon because of a knee injury resulting in a ACL rupture, for whom surgery indication for an ACL reconstruction exists and who can be operated on within three weeks after the onset of the ACL rupture.

Intervention:

n=48 patients will participate in the current study. Patients will be assigned to a suture repair of the ruptured vkb complemented by a dynamic intraligamentary stabilization (DIS) and microfracture of the femoral notch or the gold standard, a ACL reconstruction.

Primary study parameters/outcome of the study:

Self-reported functional outcome at one-year follow post surgery measured by the IKDC 2000 subjective scale.

Secundary study parameters/outcome of the study (if applicable):

Secondaire eindpunten: Self-reported functional outcome at one-year follow post surgery measured by the IKDC 2000 subjective scale 6 weeks, 3,6 and 9 months, 2,5 and 10 years post surgery, self-reported disabilities (KOOS), level of physical activity (Tegner), satisfaction (VAS) as well as IKDC physical examination (clinimetretrics) 6 weeks, 3, 6 en 9 months, 1, 2, 5 and 10 years post surgery; instrumented anteroposterior laxity, leg symmetry index for jump tests as well as isokinetic quadriceps en hamstrings force 6 en 9 months, 1, 2, 5 en 10 years after surgery; radiologic signs of arthrosis 1,2 5 and 10 years post surgery; reruptures of the ACL within 10 years post surgery, classification rupture pattern peroperative.

ELIGIBILITY:
Inclusion Criteria:

* Sportive, active patient (Tegner score =/>5)
* Age above 18 untill 30 years at time of inclusion
* Primary rupture of the anterior cruciate ligament, evidence by history (acute trauma, clicking sensation, swelling within a few hours, instability) and physical examination (positive Lachman, anterior drawer test and/or Pivot shift)
* Primary rupture indicated by MRI
* No associated ligamentuous disorde of the knee, evidenced by history, physical examination, x-ray or MRI)
* Time span between anterior cruciate ligament rupture and operation no longer than 21 days
* Willingness to comply to advised rehabilitation protocol supervised by (NFVS registrated) sports physiotherapist

Exclusion Criteria:

* Infection
* Known hypersensitive response for materials used (Cobalt, chroom, nickel)
* Serieus pre-existing malaligment of leg indicated for surgery
* Tendency for excessive scar tisseu formation, such as arthrofibrosis
* History of previous surgery on leg indicated for surgery
* History of removal of tendon on leg indicated for surgery
* Muscular, neurological or vascular disorders negatively affecting healing or rehabilitation
* Cartilage injury requiring (some kind of) cartilage repair surgery (such as microfracture or cell therapy)
* Arthrosis more dan ICRS grade 2 evidenced by x-ray
* Long(er) term use of relevant medication, such as prednisolon or cytostatica
* Pregnancy
* Know osteoporosis

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
IKDC 2000 subjective knee evaluation form | baseline, 12 months post surgery
  questionniare/self-reported functional limitations in activitities of daily living and/or sports activities

SECONDARY OUTCOMES:
IKDC 2000 subjective knee evaluation form | baseline, 6 weeks, 3-6-9-12 months, 2-5-10 years post surgery
  questionnaire/self-reported functional limitations in activitities of daily living and/or sports
IKDC 2000 objective knee evaluation form | baseline, 6 weeks, 3-6-9-12 months, 2-5-10 years post surgery
  knee physical examination form / clinimetrics
Knee Injury and Osteoarthritis Outcome Score (KOOS) | baseline, 6 weeks, 3-6-9-12 months, 2-5-10 years post surgery
  questionnaire designed to assess short and long term patient-related ouctome following knee injury on pain, symptoms, activities of daily living, sport and recreation, knee-related quality of life
Tegner Activity Level Scale | baseline, 6 weeks, 3-6-9-12 months, 2-5-10 years post surgery
  Rating scale to determine the type and intensity of sports/activities
Instrumented anteroposterior laxity | baseline, 6 weeks, 3-6-9-12 months, 2-5-10 years post surgery
LSI jump-force testing | 6-9-12 months, 2-5-10 years post surgery
  leg symmetry index for jump tests as well as isokinetic quadriceps and hamstring force tests

OTHER OUTCOMES:
Reinjuries | up till 10 years post surgery
  reinjuries or reruptures of the knee
workability | baseline, 6 weeks, 3-6-9-12 months, 2-5-10 years post surgery
  questionnaire to assess the patient's workability due to knee injury/knee surgery in order to be able to make an estimation of costs benefits between study arms
Classification of type of rupture of the ACL | during surgery
  The surgeon's opinion regarding the classification of the type of rupture of the ACL peroperative.
Complications associated with knee surgery and/or rehabilitation | baseline, 6 weeks, 3-6-9-12 months, 2-5-10 years post surgery
  The complications that occur as a result of the ACL surgery and/or rehabilitation in time.
x-ray knee | 5 and 10 years post surgery
  x-ray will be taken of the knee in order to be able to determine the degree of arthrosis

CONTACTS AND LOCATIONS:
Overall Officials: R.A.G Hoogeslag, MD, Principal Investigator — OCON
Locations (1):
- Orthopedisch Centrum Oost Nederland /ZGT, Hengelo, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
to be determined yet

REFERENCES:
- [Derived] Hoogeslag RAG, Brouwer RW, Boer BC, de Vries AJ, Huis In 't Veld R. Acute Anterior Cruciate Ligament Rupture: Repair or Reconstruction? Two-Year Results of a Randomized Controlled Clinical Trial. Am J Sports Med. 2019 Mar;47(3):567-577. doi: 10.1177/0363546519825878. PMID 30822124
- [Derived] Boer BC, Hoogeslag RAG, Brouwer RW, Demmer A, Huis In 't Veld RMHA. Self-reported functional recovery after reconstruction versus repair in acute anterior cruciate ligament rupture (ROTOR): a randomized controlled clinical trial. BMC Musculoskelet Disord. 2018 Apr 20;19(1):127. doi: 10.1186/s12891-018-2028-4. PMID 29678170